CLINICAL TRIAL: NCT07043179
Title: Comparison of Corticosteroid Injection, Nighttime Splinting, or Their Combination for Initial Treatment of Moderate-to-Severe Carpal Tunnel Syndrome: A Pragmatic, Three-Armed, Open-Label, Multicenter, Randomized Clinical Trial
Brief Title: Comparison of Corticosteroid Injection, Nighttime Splinting, or Their Combination for Initial Treatment of Moderate-to-Severe Carpal Tunnel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yun Qian (Other)
Collaborators: Shanghai 6th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Yun Qian, Principal Investigator, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-097
Record Dates: First submitted 2025-06-22; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Carpal Tunnel Syndrome (CTS)
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nighttime splinting (Other): Wear a wrist neutral position splint at night for 6 weeks as the initial treatment.
  Interventions: Device: Nighttime Splinting; Other: Evaluation and Dynamic Adjustment
- Corticosteroid injection (Other): Local corticosteroid injection (triamcinolone acetonide 40mg) as the initial treatment.
  Interventions: Drug: Corticosteroid Injection; Other: Evaluation and Dynamic Adjustment
- Combination (Other): Nighttime splinting for 6 weeks combined with local corticosteroid injection (triamcinolone acetonide 40mg) as the initial treatment.
  Interventions: Device: Nighttime Splinting; Drug: Corticosteroid Injection; Other: Evaluation and Dynamic Adjustment

INTERVENTIONS:
Device: Nighttime Splinting — Nighttime splinting for 6 weeks.
  Other Names: Wrist Splint
  Arms: Combination; Nighttime splinting
Drug: Corticosteroid Injection — Local corticosteroid injection (triamcinolone acetonide 40mg). A single injection of triamcinolone acetonide 40mg mixed with an equal volume of 1% lidocaine is administered. The injection is performed under ultrasound guidance and anatomical landmarks to target the proximal carpal tunnel. With the wrist extended, the needle is typically inserted on the ulnar side of the palmaris longus tendon, approximately 1 cm proximal to the wrist crease. If blood is aspirated or the patient reports paresthesia (which usually indicates nerve irritation), the injection site should be adjusted.
  Other Names: Steroid Injection
  Arms: Combination; Corticosteroid injection
Other: Evaluation and Dynamic Adjustment — 6 weeks later, all patients will undergo evaluation of their initial treatment. Further therapeutic decisions will be made based on physician assessment, including: continuing nighttime splinting, administering corticosteroid injections to patients who initially received only the splint, adding nighttime splinting for patients initially received only corticosteroid injections, and transitioning from nighttime splint use to continuous wear. Subsequently, evaluations will be conducted every 6 weeks, with dynamic adjustments to the treatment plan. Corticosteroid injections will be administered at least 24 weeks apart, and the second injection dosage may be adjusted based on the patient's condition, with a maximum dose of 80mg. Throughout the study period, physicians will perform electrophysiological examinations according to changes in patients' clinical status.

SUMMARY:
The goal of this clinical trial is to compare the efficacy of corticosteroid injection, night splinting, and their combined use as initial treatments for adults with moderate to severe carpal tunnel syndrome (CTS), and to assess the safety and tolerability of these interventions. The primary research questions include:

* Doe corticosteroid injection, night splinting, and their combined use as initial treatments reduce the need for surgery in participants with moderate to severe CTS?
* How do these interventions affect the improvement of patient symptoms?

Participants will:

* Receive corticosteroid injection, night splinting, or their combination as initial treatments.
* Visit the clinic once every 6 weeks over a period of one year for assessments and dynamic adjustment of the treatment plan.
* Undergo periodic assessments of wrist function, quality of life, and sleep quality using standardized questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged no less than 18 years old with idiopathic carpal tunnel syndrome of the target side diagnosed by a specialist according to the Katz diagnostic criteria;
2. The current episode has occurred within 6 weeks without treatment before eligibility assessment, and the target side has moderate-to-severe symptoms.

Exclusion Criteria:

1. Patients who have plan for surgical treatment on his or her CTS within the following 6 months;
2. Any secodary CTS caused by comorbid diseases, including rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, CPPD (calcium pyrophosphate dihydrate deposition disease), etc.;
3. History of fracture or surgery on the target side of the wrist;
4. Bilateral CTS with moderate or severe symptoms in both hands;
5. Received corticosteroid injections in the wrist within the past 6 months;
6. Patients who are unable to wear a splint due to trauma or other reasons;
7. Patients with clinical manifestations or electrophysiological changes indicative of significant axonal loss or denervation, including thenar muscle atrophy, sensory loss (two-point discrimination greater than 8 mm), absence of SNAP (sensory nerve action potential), absence of CMAP (compound muscle action potential) in the thenar muscles, etc.;
8. Patients who require long-term use of any form of analgesic medication, such as NSAIDs (nonsteroidal anti-inflammatory drugs), opioids, acetaminophen, etc.;
9. Patients who have used NSAIDs, opioids (e.g., tramadol), neuropathic pain medications (gabapentin, pregabalin, etc.), or oral corticosteroids within the past 2 weeks;
10. Patients who have received non-recommended wrist injection treatments (e.g., 5% glucose, platelet-rich plasma, ozone, chitosan, hyaluronic acid, etc.) within the past 6 months;
11. Patients who have undergone non-recommended physical therapies (e.g., electrotherapy, magnetotherapy, laser therapy, etc.) within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Surgical rate within 52 weeks | 52 weeks
  Participants will be asked if they have undergone surgery for carpal tunnel syndrome in the last 52 weeks.

SECONDARY OUTCOMES:
Change from baseline in BCTQ symptom severity subscale | 0,6,12,24,52 weeks
  Change from baseline in the score of the BCTQ symptom severity subscale (Boston Carpal Tunnel Questionnaire Symptom Severity subscale) will be compared between treatment groups at 6 ,12, 24 and 52 weeks follow-up.
Change from baseline in BCTQ function status subscale | 0,6,12,24,52 weeks
  Change from baseline in the score of the BCTQ function status subscale (Boston Carpal Tunnel Questionnaire Function Status Subscale) will be compared between treatment groups at 6 ,12, 24 and 52 weeks follow-up.
Change from baseline of EQ-VAS | 0,6,12,24,52 weeks
  The EQ-VAS is a measure of the overall health of respondents on the day of the survey. Change from baseline in the score of EQ-VAS will be compared between treatment groups at 6 ,12, 24 and 52 weeks follow-up.
Change from baseline of PSQI | 0,6,12,24,52 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality. Change from baseline in the score of the PSQI will be compared between treatment groups at 6 ,12, 24 and 52 weeks follow-up.
Change from baseline of the cross-sectional area of the median nerve | 0,52 weeks
  The median nerve cross-sectional area will be measured with musculoskeletal ultrasound. Change from baseline of the cross-sectional area will be compared at 52 weeks follow-up.
The incidence rate of clinical and electrophysiological changes indicative of new-onset axonal loss or denervation within 52 weeks | 52 weeks
  Researchers will assess and record whether there are any new clinical or electrophysiological changes indicating axonal loss or denervation during follow-up. The incidence rates of these changes in different treatment groups will be compared at the 52-week follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Jinjiang Municipal Hospital(Shanghai Sixth People's Hospital Fujian Campus), Jinjiang, Fujian
  - Yancheng Third People's Hospital, Yancheng, Jiangsu
  - Shanghai Sixth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study for publication, by reasonable request via email to the corresponding author.